CLINICAL TRIAL: NCT06575972
Title: A Clinical Study to Assess the Effects of JoyRise Recovery Powder on Mitigating Alcohol Aftereffects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joyrise (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20374
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Aftereffects; Anxiety; Cognitive Impairment
Keywords: Cognitive Function; Hangover; Anxiety Reduction
MeSH Terms: conditions — Anxiety Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy of JoyRise Recovery Powder in mitigating the aftereffects of alcohol consumption. The study involves two groups: one receiving the active supplement (JoyRise Recovery Powder) and the other receiving a placebo.
Who Masked: Participant, Investigator
Masking Description: This study uses a double-blind design, meaning that both the participants and the investigators are unaware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JoyRise Recovery Powder (Experimental): Participants in this arm will receive JoyRise Recovery Powder, a dietary supplement containing Dihydromyricetin (DHM) and other natural ingredients.
  Interventions: Dietary Supplement: JoyRise Recovery Powder
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo solution that is visually and tastefully similar to the JoyRise Recovery Powder but contains no active ingredients.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: JoyRise Recovery Powder — JoyRise Recovery Powder is a dietary supplement that contains Dihydromyricetin (DHM) and other natural ingredients. It is designed to mitigate the aftereffects of alcohol consumption. Participants will mix one serving in 8-12 oz of water and consume it the morning after alcohol consumption.
  Arms: JoyRise Recovery Powder
Dietary Supplement: Placebo — A placebo solution that is visually and tastefully similar to JoyRise Recovery Powder but contains no active ingredients. It will be mixed in 8-12 oz of water and consumed the morning after alcohol consumption.
  Arms: Placebo

SUMMARY:
This study assesses the effectiveness of JoyRise Recovery Powder in reducing alcohol aftereffects, cognitive impairment, and anxiousness among participants aged 35-54 who consume alcohol. Participants will be randomly assigned to either the JoyRise group or a placebo group. The study will measure hangover symptoms, cognitive function, and overall well-being through a series of questionnaires and cognitive tests at baseline, 30 minutes after product consumption, and 4 hours later.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-54, male or female
* Regular alcohol consumption
* Event planned within one month that involves alcohol consumption
* Willingness to avoid new medications or supplements during the study period
* Must confirm that they will not drive while under the influence of alcohol.

Exclusion Criteria:

* Anyone not in good health.
* Anyone who has any chronic health conditions such as oncological or psychiatric disorders.
* Anyone who has any known serious allergic reactions that require the use of an Epi-Pen.
* Anyone who is pregnant, breastfeeding, or trying to conceive.
* Anyone who cannot/ will not commit to the study protocol.
* Anyone with a history of substance abuse.
* Anyone who has undergone an invasive medical procedure in the six months prior to the study, or has a procedure planned during the study duration.
* Anyone currently using any medications that may affect their response to alcohol or impact hangover symptoms, such as diuretics (water pills) or medication for hypertension.
* History of severe reactions or sensitivity to alcohol.
* Anyone currently taking glutathione.

Ages: 35 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Symptoms Associated with Alcohol Aftereffects | Baseline and 30 minutes after product consumption on the day following alcohol consumption.
  Measurement of the reduction in alcohol aftereffects using the Alcohol Hangover Questionnaire (AHQ). Participants will self-report their symptoms, such as headache, nausea, and tiredness.

SECONDARY OUTCOMES:
Improvement in Cognitive Function | Baseline and 30 minutes after product consumption on the day following alcohol consumption.
  Measurement of cognitive function using Double Trouble (which assesses selective attention and processing speed). Participants will complete this assessment to determine any changes in cognitive function.
Improvement in Cognitive Function | Baseline and 30 minutes after product consumption on the day following alcohol consumption.
  Measurement of cognitive function using two cognitive tests: Feature Match (which assesses focus and processing). Participants will complete this assessment to determine any changes in cognitive function.
Reduction in Feelings of Anxiousness | Baseline and 30 minutes after product consumption on the day following alcohol consumption.
  Measurement of reduction in feelings of anxiousness using self-reported questionnaires. Participants will rate their anxiety levels to determine if the product provides a calming effect.
Increased User Satisfaction with Overall Well-being | Baseline and 4+ hours after product consumption on the day following alcohol consumption.
  Measurement of user satisfaction with overall well-being through self-reported questionnaires. Participants will rate their satisfaction with their physical and mental state post-alcohol consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No